CLINICAL TRIAL: NCT02485756
Title: An Educational Intervention to Increase Knowledge of Drug-drug Interactions Between Antiepileptics and Hormonal Contraception Among Reproductive-aged Women With Epilepsy.
Brief Title: Counseling on the Interaction of Hormonal Contraceptives and Antiepileptics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Sheila Mody, Associate Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UCSD130139
Record Dates: First submitted 2013-09-26; First posted 2015-06-30 (Estimated); Last update posted 2019-06-07 (Actual); Status verified 2019-06

CONDITIONS: Epilepsy
Keywords: Drug interactions
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Educational handout (Experimental): Participants in the intervention group will read an educational handout on hormonal contraceptives/antiepileptic interactions.
  Interventions: Other: Educational handout
- Control (no educational handout) (No Intervention): Those in the standard care group will not receive the educational handout.

INTERVENTIONS:
Other: Educational handout — Topics include: interactions between AED and certain hormonal contraceptives, Center for Disease Control and Prevention (CDC) recommendations for alternative contraceptive methods that are not known to interact with AEDs, contraceptive failure rates
  Arms: Educational handout

SUMMARY:
Previous studies have shown that women on anti-seizure medications are not informed about the pharmaceutical drug interactions between anti-seizure medications (antiepileptic drugs, AEDs) and certain hormonal contraceptive. The goal of this proposed study is to develop and assess the efficacy of an educational handout for participants on the ways AEDs and certain hormonal contraceptives can interact to alter effectiveness of the medications. Reproductive age women (18-45 years old) will be recruited from UCSD Health System Epilepsy clinics. If a patient agrees to participate, she will be given a knowledge exam prior to the clinic appointment to establish baseline understanding of hormonal contraceptive and AED interactions and then the participant will be randomized to receive the intervention (educational handout) or the standard of care (no educational handout). Those in participants in the intervention group will read an educational handout on hormonal contraceptives/AED interactions. Those in the standard care group will not receive this handout and the same knowledge exam will be re-administered to all of the participants after they have completed their appointments to check for knowledge comprehension and short-term knowledge retention. A same-day post-test questionnaire will evaluate participant's intention to discuss hormonal contraceptives/AED interactions with their gynecologist, neurologist or primary care physician.

ELIGIBILITY:
Inclusion Criteria:

* Age of participants: 18-45 years old
* Gender of participants: Female
* Ethnic Background: No limitation, will include minorities
* Health Status: on at least one antiepileptic medication
* Sexually active with men
* English speaking

Exclusion Criteria:

* Currently Pregnant
* History of hysterectomy or sterilization procedure
* Removal of both ovaries
* Cannot read or comprehend English language
* Unable to provide informed consent
* Attempting to become pregnant
* Not sexually active with men
* No active telephone number for follow-up contact

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Score on 10 question test | Score on pretest (prior to intervention/standard care) and post-test (after intervention/standard care).
  Change in score on knowledge examination (comparison of pretest and posttest score)

CONTACTS AND LOCATIONS:
Overall Officials: Sheila Mody, MD, Principal Investigator — UC San Diego; Marisa Hildebrand, MPH, Study Director — UCSD
Locations (1):
- UC San Diego Medical Center, San Diego, California, United States

REFERENCES:
- [Derived] Mody SK, Haunschild C, Farala JP, Honerkamp-Smith G, Hur V, Kansal L. An educational intervention on drug interactions and contraceptive options for epilepsy patients: a pilot randomized controlled trial. Contraception. 2016 Jan;93(1):77-80. doi: 10.1016/j.contraception.2015.07.008. Epub 2015 Jul 18. PMID 26197260